CLINICAL TRIAL: NCT04786587
Title: Evaluation of the Diagnostic Value of the Self-report T-ACE for Screening of High-risk Alcohol Consumption During Pregnancy : Comparison With the Dosage of a Blood Biomarker Used as Gold Standard. AUTOQUEST Study.
Brief Title: Alcohol Self-reporting During Pregnancy. AUTOQUEST Study.
Acronym: AUTOQUEST
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Other Study IDs: 2018_85; 2021-A00058-33 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2021-03-04; First posted 2021-03-08 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-03

CONDITIONS: Alcohol Drinking; Pregnancy
Keywords: screening; alcohol consumption; pregnancy; self report
MeSH Terms: conditions — Alcohol Drinking | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pregnant woman
  Interventions: Diagnostic Test: blood test; Other: self-administered questionnaire

INTERVENTIONS:
Diagnostic Test: blood test — Each pregnant woman completes the self-report during her prenatal consultation and will have a unique blood sampling for dosage of phosphatidylethanol after she returned her self-report to the practitioner and if she is included in the study (informed consent given).
  the blood test for dosage of phosphatidylethanol will be offered to all eligible pregnant women in each maternity clinic of the study during the recruitment period. There will not be different arms in this study.
Other: self-administered questionnaire — Each pregnant woman completes the self-report during her prenatal consultation and will have a unique blood sampling for dosage of phosphatidylethanol after she returned her self-report to the practitioner and if she is included in the study (informed consent given).
  A self-report, including the T-ACE, is the usual prenatal consultation procedure in the three maternities of the study. The specific procedure for the study is to perform a blood test for dosage of phosphatidylethanol in eligible pregnant women after informed consent.

SUMMARY:
The effects of alcohol consumption during pregnancy have been known for decades. However, alcohol consumption in pregnant women remains today a public health problem and its identification is primordial. During pregnancy, standardized self-reports such as T-ACE would help identify early women with high-risk alcohol consumption. T-ACE appears to be one of the most used during pregnancy but its diagnostic value is not objectively known.

To evaluate the diagnostic value of T-ACE self-report in the detection of high-risk alcohol consumption during pregnancy, by comparison with the dosage of a biomarker in blood.

Material and methods Multicentric diagnostic prospective study of 2425 pregnant women followed in 3 hospitals of North of France. The self-report will be offered to all women during their prenatal consultation in these 3 maternity clinics. When they returned their self-report to the medical practitioner, a unique blood test of phosphatidylethanol will be proposed to them for a period of one year. Made after informed consent, this dosage will be used as a gold standard of an alcohol consumption during the previous three weeks to establish the diagnostic value of T-ACE. An alcohol consumption will be considered " at high risk " if blood phosphatidylethanol is ≥ 20 µg/L.

With a predictable 25% rejection rate and a positive 4% T-ACE frequency, the inclusion of 2425 patients should permit to estimate sensitivity, specificity, positive predictive value (PPV) and negative predictive value (NPV) of T-ACE with a satisfactory 95% confidence interval in this population.

The evidence of a link between positive T-ACE and real high-risk alcohol consumption in pregnant women would objectively validate the use of this self-report during pregnancy.

The T-ACE within the self-report (self-administered questionnaire) set up in these 3 maternity hospitals in the North of France is already a reference thanks to its several advantages to better identify psychosocial risk situations and especially high-risk alcohol consumption during pregnancy than medical history. If T-ACE appeared to be a sensitive and specific method for identifying high-risk alcohol use during pregnancy, it could be generalized in the follow-up of pregnant women in our country.

ELIGIBILITY:
Inclusion Criteria:

* pregnant woman over 18 years old, presenting in one of the three maternities of the study for her prenatal care
* and having returned her self-report
* and having given her written consent
* no exclusion criteria

Exclusion Criteria:

* woman under 18 years old
* or not pregnant
* or not having returned her self-report
* or woman who refused to participate in the study (absence of written consent)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Pregnant women
Study Population: Pregnant women followed in 3 maternity hospitals in the North of France
Sampling Method: Probability Sample
Enrollment: 2425 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Calcul of sensitivity of the self-report T-ACE compared to the result of phosphatidylethanol dosage (µg/L) | At Baseline
  the calcul of sensitivity of the self-report T-ACE to detect a high-risk alcohol consumption in pregnant women, compared to the result of phosphatidylethanol dosage in blood sampling used as gold standard of an alcohol consumption during the previous three weeks
  The blood sampling for dosage of phosphatidylethanol is done when the self-report is returned to the medical practitioner by the pregnant woman, if she is included in the study after giving her informed consent.

SECONDARY OUTCOMES:
Calcul of specificity, PPV and NPV of the self-report T-ACE compared to the result of phosphatidylethanol dosage (µg/L) | At Baseline
  The calcul of specificity, PPV and NPV of the self-report T-ACE to detect a high-risk alcohol consumption in pregnant women, compared to the result of phosphatidylethanol dosage in blood sampling used as gold standard of an alcohol consumption during the previous three weeks.
  The blood sampling for dosage of phosphatidylethanol is done when the self-report is returned to the medical practitioner by the pregnant woman, if she is included in the study after giving her informed consent

CONTACTS AND LOCATIONS:
Overall Officials: Damien SUBTIL, MD,PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- University Hospital, Lille, Lille, France